CLINICAL TRIAL: NCT04868955
Title: Evaluation of Oral Screen Training With IQoro as Treatment for Dysphagia After Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Rebecca Norrman and Elin Rova (Other)
Responsible Party: Sponsor-Investigator, Rebecca Norrman and Elin Rova, Speech and language pathologists, Ostergotland County Council, Sweden
Organization: Ostergotland County Council, Sweden (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-00636
Record Dates: First submitted 2021-04-21; First posted 2021-05-03 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Stroke; Dysphagia
MeSH Terms: conditions — Stroke; Deglutition Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Usual care and oral screen (IQoro®) training.
  Interventions: Other: Oral screen training
- Control group (No Intervention): Usual care.

INTERVENTIONS:
Other: Oral screen training — Oral screen training (IQoro®) during 13 weeks.
  Arms: Intervention group

SUMMARY:
Purpose The purpose of the study is to evaluate if training with oral screen IQoro® improves swallowing in patients with dysphagia after stroke.

Method Inpatient from a stroke unit in Sweden who have been assessed with fiberoptic endoscopic evaluation of swallowing(FEES) which proves swallowing difficulties (dysphagia) were recruited. The participants were randomise to control- or intervention group. Both groups received usual care. The intervention group were instructed to oral screen (IQoro®) training for 13 weeks. Follow up with FEES was made 13 weeks post of recruitment. The assess with FEES was recorded and the recordings are going to be analyzed afterwards to compare the swallowing ability between baseline and follow up in group and between group.

ELIGIBILITY:
Inclusion Criteria:

* Inpatient at stroke unit at Vrinnevisjukhuset ward 1, due to stroke.
* Patient assessed to have dysphagia (score ≥1 on one of the studied parameters)according to FEES.
* Patient who is able to handle IQoro® according to instructions, independently or with support of assistance from relatives or staff.

Exclusion Criteria:

* Patients with dysphagia of a cause other than stroke.
* Patient with impaired cognitive skill, motor and / or language ability that prevents the possibility of performing training with IQoro®, despite possible support from assistance from relatives or staff.
* Patient who wishes training with the Muppy oral screen® related to saliva leakage.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2019-04-26 (Actual); Primary Completion 2021-05-03 (Estimated); Study Completion 2021-05-03 (Estimated)

PRIMARY OUTCOMES:
Change in swallowing function due to secretion in the pharynx. | From baseline to follow up (13 weeks after baseline).
  Changes in swallowing function based on the parameter secretion in the pharynx. Estimates from "Secretion severity rating scale", 0-3. 0= Normal rating and 3= Secretion in the laryngeal vestibule that are not cleared.
  Estimates are based on recording from FEES.
Change in swallowing function due to aspiration and penetration. | From baseline to follow up (13 weeks after baseline).
  Changes in swallowing function based on the parameters aspiration and penetration in the pharynx. Estimates from "Penetration aspiration scale", 0-8. 0= No entry of material into the larynx or trachea, 8= Materials enter the trachea with no attempt to clear.
  Estimates are based on recording from FEES.
Change in swallowing function due to residual in the pharynx. | From baseline to follow up (13 weeks after baseline).
  Change in swallowing function due to residual in the pharynx, 0-1. 0= No or a small amount of residual, 1= A pool of residual after the first swallow.
  Estimates are based on recording from FEES.

SECONDARY OUTCOMES:
The patient's experience of swallowing | From baseline to follow up (13 weeks after baseline)
  The patient estimates its own swallowing ability on the basis of a "Visual analogue scale" (VAS), 0-100. 0= No affected swallowing function and 100= Very affected swallowing function).
Change in swallowing function due to oral intake. | From baseline to follow up (13 weeks after baseline).
  Change in oral intake estimates from "Functional oral intake scale" (FOIS), 1-7. 1= Nothing by mouth, 7= Total oral diet with no restrictions.
  Estimates are based on advice the patient received regarding the oral intake.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca U Norrman, Master, Principal Investigator — Ostergotland County Council, Sweden; Elin AM Rova, Master, Principal Investigator — Ostergotland County Council, Sweden
Locations (1):
- Vrinnevisjukhuset, Norrköping, Östergötland County, Sweden

IPD SHARING:
Plan to Share IPD: No
Data will only be reported and shared at group level.